CLINICAL TRIAL: NCT03528720
Title: Evaluation System and Clinical Application for Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018188H
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Diabetic Retinopathy
Keywords: Tomography, Optical Coherence; Fluorescein Angiography; Fundus photographs
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetic retinopathy(DR) is one of the most common and serious microvascular complications of diabetes,which is the primary cause of vision loss of diabetic patients. The risk of blindness is 25 times that of healthy people.Fundus fluorescein angiography (FFA) is the gold standard for diagnosing the stage of diabetic retinopathy.However,FFA is an invasive examination which requires the patient to be in good physical condition and is not suitable for large-scale screening.Therefore, it is important to build up an evaluation system for early diagnosis of DR,which is more convenient, safer, and non-invasive.Firstly, this study will retrospectively analyze the FFA images of DR to find the earliest and most frequently occurring fundus quadrant.Secondly,based on the retrospective analysis results, a prospective comparative study will be conducted,which combines the fundus photography with optical coherence tomography angiography(angio-OCT) and physical indicators to find out whether it has consistency, sensitivity and specificity with FFA in diagnosing the stage of DR in order to build up a more effective,safer and faster evaluation system and clinical application for DR.

DETAILED DESCRIPTION:
Firstly, this study will retrospectively analyze the FFA images of DR to find the earliest and most frequently occurring fundus quadrant.Secondly,based on the retrospective analysis results, a prospective comparative study will be conducted,which combines the fundus photography with angio-OCT and physical indicators to find out whether it has consistency, sensitivity and specificity with FFA in diagnosing the stage of DR.Finally，based on all the results,to build up a more effective,safer and faster evaluation system and clinical application for DR.

ELIGIBILITY:
Inclusion Criteria:

Patients with diabetic retinopathy

Exclusion Criteria:

Refractive interstitial turbidity Cannot cooperate with examiner Retinal surgery in patients Malignant tumors Hematological diseases Immune diseases Glaucoma or other retinal diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The retrospective study needs 150 people.The prospective comparative study needs 200 people.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
The earliest and most frequently occurring fundus quadrant of diabetic retinopathy in fundus fluorescein angiography. | 2 years
  The study is to find the earliest and most frequently occurring fundus quadrant of diabetic retinopathy.Based on the the retrospective analysis results, a prospective comparative study will be conducted to build up a evaluation system and clinical application for diabetic retinopathy.We divided the FFA images into nine quadrants: posterior pole, superior, superior nasal, nasal, inferior nasal, inferior, inferior temporal, temporal, and superior temporal. The qualitative analysis of diabetic retinopathy in each quadrant was performed. The earliest and most common fundus quadrant of diabetic retinopathy was then assessed using a rank sum test, t-test, and analysis of variance.

CONTACTS AND LOCATIONS:
Locations (1):
- Qianli Meng, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Xie J, Zhang L, Cui Y, Zhang G, Wang J, Zhang A, Chen X, Huang T, Meng Q. Differential distribution of manifest lesions in diabetic retinopathy by fundus fluorescein angiography and fundus photography. BMC Ophthalmol. 2020 Dec 1;20(1):471. doi: 10.1186/s12886-020-01740-2. PMID 33261573